CLINICAL TRIAL: NCT04847999
Title: Impact of Dark Chocolate Consumption on Glucose Levels of People With Diabetes
Brief Title: Dark Chocolate and Glucose Levels in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: H20-02122
Record Dates: First submitted 2021-01-05; First posted 2021-04-19 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Chocolate bars will be identical and wrapped equally and labeled as A and B, by Ross Chocolates (prepared in the same mold and packaged identically) who are not involved in any other aspects of the study, allowing for blinding of research team and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Dark Chocolate then Ross Dark Chocolate (Experimental): A Conventional dark chocolate bar will be consumed and after a 1-week washout period, Ross Dark chocolate will be consumed.
  Interventions: Dietary Supplement: Dark chocolate
- Ross Dark Chocolate and then Conventional chocolate (Experimental): A dark chocolate bar sweetened with stevia, erythritol, and inulin - Ross Dark Chocolate will be consumed and after a 1-week washout period, Conventional Dark chocolate will be consumed.
  Interventions: Dietary Supplement: Dark chocolate

INTERVENTIONS:
Dietary Supplement: Dark chocolate — Dark chocolate

SUMMARY:
Diabetes is a growing concern in the world with an estimated 9.3% of adults, ages 20-79, with it in 2019, type 2 diabetes accounting for 90% of this total. A common recommendation for individuals with diabetes is to limit sugars and sweets as it may cause a high blood glucose response. As a result, chocolate is often avoided due to the sugar content; though, high-polyphenol chocolate may have a beneficial effect on hyperglycaemia and vascular function. The sugar-free chocolate from Ross Chocolates is formulated with a blend of inulin, erythritol, and stevia. These alternatives to sugar are not expected to cause a significant change in blood glucose levels following consumption. The main objective of this study is to verify glucose levels before and after consumption of Ross Chocolates' blend of sweeteners dark chocolate and conventional chocolate in people with diabetes.

DETAILED DESCRIPTION:
Individuals with type 1 or type 2 diabetes (10 participants each) will consume a Ross Chocolate or conventional sugar-sweetened dark chocolate bar on two occasions in a randomized crossover trial. Blood glucose levels will be measured by finger prick for 120 minutes after consumption to determine postprandial glucose excursions after consumption of each type of chocolate bar.

Due to the COVID-19 pandemic, the trial was converted to be completed remotely/virtually with participants completing the testing at their home under the supervision of a research team member who will describe the study procedures and monitor testing via video conferencing.

ELIGIBILITY:
Inclusion Criteria:

* physician-diagnosed T1D or T2D of ≥1 year;
* current HbA1c of 6.5-8.5%;
* BMI: 25-40 kg/m2;
* blood pressure of <160/99 mm Hg assessed according to guidelines;
* non-smoking;
* not on hormone replacement therapy, corticosteroids, or anti-inflammatory medications;
* 18-75 years old.

Exclusion Criteria:

* Are taking more than 2 glucose lowering medications;
* Are ongoing medical treatment for diseases such as cancer, auto-immune or inflammatory disease, liver or kidney disorders;
* Have allergy, intolerance or aversion to cocoa, stevia, erythritol, inulin, or any other dietary restrictions (e.g., vegan) that will prevent them from following the standardized study diets;
* Are unable to follow remote guidance by internet or smartphone;
* Are unable to follow the controlled diet instructions;
* Are unable to read or communicate in English.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Dark Chocolate Then Ross Dark Chocolate: Start crossover with a standard dark chocolate bar and then a a dark chocolate bar sweetened with stevia, erythritol, and inulin.
- Ross Dark Chocolate Then Conventional Dark Chocolate: Start with a dark chocolate bar sweetened with stevia, erythritol, and inulin and then a conventional dark chocolate.
Period: Overall Study
Arm/Group | Conventional Dark Chocolate Then Ross Dark Chocolate | Ross Dark Chocolate Then Conventional Dark Chocolate
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants with type 1 and type 2 diabetes included for 2 crossover conditions: Ross chocolate and then Conventional chocolate or Conventional chocolate and then Ross chocolate.
Groups:
- All Study Participants: Participants with type 1 and type 2 diabetes completed this crossover study consuming either a conventional dark chocolate and then Ross dark chocolate OR Ross dark chocolate and then conventional dark chocolate.
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  Canada | 13
Body mass [Mean (Standard Deviation); unit: kg] | 84.9 (23.3)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 29.0 (5.6)
HbA1c [Mean (Standard Deviation); unit: %] | 7.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Incremental Area Under the Curve
Description: A self-monitoring blood glucose device (OneTouch Verio IQ® kit Blood glucose monitoring system) will be used to measure blood glucose levels before and after consumption of chocolates. Incremental area under the curve will calculate the glucose above baseline fasting values across 120 minutes.
Time Frame: 0 and 120 min after consumption of chocolate bar
Population: People with Type 1 and Type 2 diabetes
Measure: Mean (Standard Error); unit: mM x 120 minutes
Groups:
- Dark Chocolate: Conventional Dark chocolate
- Ross Dark Chocolate: sugar-free dark chocolate
Arm/Group | Dark Chocolate | Ross Dark Chocolate
Number analyzed (Participants) | 13 | 13
mM x 120 minutes | 240.5 (55.81) | 83.81 (46.18)

2. Secondary Outcome: Peak Blood Glucose Concentration
Description: Highest blood glucose value measured after consumption of the chocolate bar
Time Frame: 0 and 120 minutes after consumption of chocolate bar
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Ross Dark Chocolate: All participants in the Ross dark chocolate condition
- Conventional Dark Chocolate: All participants in the Conventional dark chocolate condition
Arm/Group | Ross Dark Chocolate | Conventional Dark Chocolate
Number analyzed (Participants) | 13 | 13
mmol/L | 10.6 (2.9) | 11.9 (4.1)

3. Secondary Outcome: Peak Blood Glucose Concentration Above Baseline
Description: Highest blood glucose value above fasting baseline after consumption of the chocolate bar
Time Frame: Throughout study completion: 0-120 minutes after consumption of chocolate bar
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ross Dark Chocolate | Conventional Dark Chocolate
Number analyzed (Participants) | 13 | 13
mmol/L | 2.2 (2.2) | 3.5 (2.9)

4. Secondary Outcome: Blood Glucose
Description: A self-monitoring blood glucose device (OneTouch Verio IQ® kit Blood glucose monitoring system) will be used to measure blood glucose levels before and after consumption of chocolates. Total area under the curve will calculate the glucose above zero across 120 minutes.
Time Frame: 0 and 120 minutes
Measure: Mean (Standard Deviation); unit: mmol x 120min
Arm/Group | Ross Dark Chocolate | Conventional Dark Chocolate
Number analyzed (Participants) | 13 | 13
mmol x 120min | 1090.8 (257.7) | 1247.5 (390.1)

5. Other Pre Specified Outcome: Taste Questionnaire - 0 to 100 Point Scale
Description: Self-reported taste of chocolate bars will be assessed by questionnaire with ratings from awful (0), average (50) to fantastic (100).
Time Frame: Throughout study completion:120 min after consumption of chocolate bar
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ross Dark Chocolate | Conventional Dark Chocolate
Number analyzed (Participants) | 13 | 13
score on a scale | 51.6 (22) | 66 (18.5)

ADVERSE EVENTS:
Time Frame: Duration of intervention period with an average of 2 weeks.
Groups:
- Conventional Dark Chocolate and Then Ross Dark Chocolate: Participants consuming a conventional dark chocolate and then Ross dark chocolate.
- Ross Dark Chocolate and Then Conventional Dark Chocolate: Participants consuming Ross dark chocolate and then conventional dark chocolate.
Arm/Group | Conventional Dark Chocolate and Then Ross Dark Chocolate | Ross Dark Chocolate and Then Conventional Dark Chocolate
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
Limitations include small number of subjects recruited and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT04847999/Prot_SAP_000.pdf